CLINICAL TRIAL: NCT00717327
Title: Medication Reconciliation List and Adolescent Functional Health Literacy
Brief Title: Adolescent Knowledge of Their Medications
Status: Completed | Type: Observational
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Dr. Kasi M. Chu, Brooke Army Medical Center Adolescent Clinic
Other Study IDs: C.2008.155
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Subjects' Understanding of Prescribed Medications
Keywords: MRL; Adolescents; Health Literacy
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Counseling for subjects who do not know their medications — Physician interviewer will provide counseling to subjects who indicate through answers that they do not know their medication names.

SUMMARY:
Do adolescents know about their medications?

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 12 and 23 who are able to answer questions regarding their prescribed medications (no receptive or expressive disability)

Exclusion Criteria:

* Adolescents outside age range of 12 and 23 who have receptive and/or expressive disability

Ages: 12 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents enrolled in an primary care clinc.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Subjects' ability to identify name and purpose of medication. | Clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Chistopher C Dillon, MD, Study Director — Brooke Army Medical Center Adolescent Clinic
Locations (1):
- Brooke Army Medical Center Adolescent Clinic, San Antonio, Texas, United States